CLINICAL TRIAL: NCT01698801
Title: A Phase 2, Multicenter, Open-label, Single Arm Study of Lenalidomide (CC-5013) in Combination With Low-dose Dexamethasone in Japanese Patients With Previously Untreated Multiple Myeloma
Brief Title: A Phase 2 Study of Lenalidomide to Evaluate the Efficacy in Japanese Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-025
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Multiple Myeloma
Keywords: Lenalidomide; dexamethasone; newly diagnosed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide plus dexamethasone (Experimental): Lenalidomide plus low-dose dexamethasone
  Interventions: Drug: Lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — 25 mg oral lenalidomide once daily on Days 1-21 of each 28-day cycle
  Other Names: Revlimid
Drug: dexamethasone — 40 mg oral dexamethasone once daily on Days 1, 8, 15 and 22 of each 28-day cycle
  Other Names: LenaDex

SUMMARY:
To determine the efficacy of lenalidomide in combination with low-dose dexamethasone in Japanese subjects with previously untreated multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years at the time of signing the informed consent document
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted
* Able to adhere to the study visit schedule and other protocol requirements
* Previously untreated, symptomatic multiple myeloma
* Have measurable disease by protein electrophoresis analyses
* At least 65 years of age or older or, if younger than 65 years of age, not candidates for hematopoietic stem cell transplantation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Must agree to comply to Lenalidomide Pregnancy Prevention Risk Management Plan

Exclusion Criteria:

* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Any condition that confounds the ability to interpret data from the study
* Previous treatment with anti-myeloma therapy
* Pregnant or lactating females
* Any of the following laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 1,000/microL (1.0 × 10^9/L )
  * Untransfused platelet count (a platelet count drawn at least 7 days after the administration of the last platelet transfusion) < 50,000 cells/microL (50 × 10^9/L)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3.0 × upper limit of normal
* Renal failure requiring hemodialysis or peritoneal dialysis
* Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years
* Subjects who are unable or unwilling to undergo antithrombotic therapy.
* Peripheral neuropathy of ≥ grade 2 severity.
* Uncontrolled systemic fungal, bacterial, or viral infection
* Known human immunodeficiency virus (HIV) positivity (subjects who are receiving antiretroviral therapy for HIV disease)
* Hepatitis Bs (HBs) antigen-positive, or hepatitis C virus (HCV) antibody-positive. In case HBc antibody and/or HBs antibody is positive even if HBs antigen-negative, a Hepatitis B virus (HBV) DNA test should be performed and if positive the subject will be excluded.
* Primary AL (immunoglobulin light chain) amyloidosis and myeloma complicated by amyloidosis.
* Ineligible for dexamethasone or dexamethasone is contraindicated.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2013-11-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Study Director — Celgene K.K.
Locations (24):
- Japan (24):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Kameda Medical Center, Kamogawa, Chiba
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Ehime University Hospital, Touon, Ehime
  - Nishigunma National Hospital, Shibukawa, Gunma
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Iwate Medical University, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kinki University Hospital, Faculty of Medicine, Sayama, Osaka
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - National Disaster Medical Center, Tachikawa, Tokyo
  - Kagoshima Medical Center, Kagoshima
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Niigata Cancer Center Hospital, Niigata
  - Okayama Medical Center, Okayama
  - Osaka Red Cross Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
  - Keio University Hospital, Tokyo

REFERENCES:
- [Result] Suzuki K, Shinagawa A, Uchida T, Taniwaki M, Hirata H, Ishizawa K, Matsue K, Ogawa Y, Shimizu T, Otsuka M, Matsumoto M, Iida S, Terui Y, Matsumura I, Ikeda T, Takezako N, Ogaki Y, Midorikawa S, Houck V, Ervin-Haynes A, Chou T. Lenalidomide and low-dose dexamethasone in Japanese patients with newly diagnosed multiple myeloma: A phase II study. Cancer Sci. 2016 May;107(5):653-8. doi: 10.1111/cas.12916. Epub 2016 Mar 30. PMID 26914369

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an ongoing open-label, single arm, 5 year study consisting of a 28-day screening period followed by a treatment period where participants receive lenalidomide and dexamethasone until their disease progresses or the lenalidomide is discontinued for any reason. This report includes data up to the cut-off of 15 July 2014.
Groups:
- Lenalidomide Plus Dexamethasone: Lenalidomide 25 mg orally once daily for 21 days in each 28-day cycle until progressive disease or lenalidomide discontinuation for any reason.
  Dexamethasone 40 mg orally once daily on Days 1, 8, 15 and 22 in each 28-day cycle until progressive disease or lenalidomide discontinuation for any reason.
Period: Treatment Phase
Arm/Group | Lenalidomide Plus Dexamethasone
Started | 26
Completed | 15 (Completed includes participants who continued to receive study medication and treatment is ongoing.)
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 1
Not completed — Other | 4
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression | 1
Period: Follow Up Phase
Arm/Group | Lenalidomide Plus Dexamethasone
Started | 11 (11 participants did not complete the study and moved into the follow up phase lasting up to 5 years.)
Completed | 6 (Completed includes participants who remain in follow-up for up to 5 years from start of treatment)
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of all participants enrolled independent of whether they received study treatment or not.
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (7.01)
Age, Customized [Number; unit: participants]
  ≤ 75 Years Old | 14
  > 75 Years Old | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Multiple Myeloma Stage before Study Entry [Number; unit: participants] — The International Staging System (ISS) divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels.
  Stage I: Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is above 3.5 (g/L);
  Stage II: Neither stage I or III, meaning that either:
  * The beta-2 microglobulin level is between 3.5 and 5.5 (with any albumin level), OR
  * The albumin is below 3.5 while the beta-2 microglobulin is less than 3.5
  Stage III: Serum beta-2 microglobulin is greater than 5.5.
  participants
    Stage I | 7
    Stage II | 14
    Stage III | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = Fully Active | 13
    1= Restrictive but Ambulatory | 7
    2 = Ambulatory but Unable to Work | 6
    3 = Limited Self-Care | 0
    4 = Completely Disabled | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Number of Complete Responses (CR) plus Very Good Partial Response (VGPR) plus Partial Response (PR) based on the International Myeloma Working Group criteria (IMWG). Any participant who achieved a CR, VGPR, or PR while on study treatment was defined as a responder.
  CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From first dose until the data cut-off date of 15 July 2014. Median time on follow-up was 61.6 weeks.
Population: Efficacy Evaluable (EE) Population consists of all participants who met the protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 24
percentage of participants | 87.5
Statistical Analysis 1: Comparison: Lenalidomide Plus Dexamethasone; Test type: Superiority or Other; p < 0.0001, Binomial test for dichotomized response — One sample binomial test for the overall response rate was performed to provide p-value (significance level: 0.05) based on EE population. The hypotheses of interest are: H0: p = 0.3, H1: p ≠ 0.3, where p is overall response; Overall dichotomized response rate = 87.5, 95% CI 2-sided [74.269 to 100]

2. Secondary Outcome: Time to Response
Description: Time to response was calculated for the responders as the time from the first dose date to the initial documented response (CR, VGPR or PR).
  CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. If present at baseline a ≥ 50% reduction in size of soft tissue plasmacytomas is also required.
Time Frame: From the first dose of study drug treatment until the data cut-off date of 15 July 2014. Median follow-up time was 61.6 weeks.
Population: Efficacy Evaluable (EE) Population consists of all participants who meet protocol requirements (all eligibility criteria) and were evaluated after receiving at least one dose of study drug
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 24
months | 1.97 [0.9 to 13.8]

3. Secondary Outcome: Duration of Response
Description: Duration of response was calculated for the responders as the time from the initial documented response (CR or VGPR or PR) to the first documented progression or death due to any cause, whichever occurred first. Duration of response for participants last known to be alive with no progression after a CR, VGPR, or PR were censored at the date of last adequate response assessment.
Time Frame: From the first dose of study drug treatment until the data cut-off date of 15 July2014. Median follow up time was 61.6 weeks.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 21
months | NA [10.550 to NA] — The median duration of response based on Kaplan-Meier estimate had not been reached by the 15 July 2014 data cut-off date.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated as the time from the first dose date to the first documented progression based on IWG criteria or death due to any cause, whichever occurred first. If progression or death was not documented at the time of data cutoff date, these observations were censored at the last adequate assessment date showing evidence of no progression or death.
Time Frame: From the first dose of study drug treatment until the data cut-off date of 15 July 2014. Median follow-up for PFS assessments was 61.6 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 24
months | NA [NA to NA] — The median time to progression free survival based on Kaplan-Meier estimate had not been reached by the 15 July 2014 data cut-off date.

5. Secondary Outcome: Overall Survival (OS)
Description: The time from the start of study treatment to death due to any cause. OS was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: From the first dose of study drug treatment until the data cut-off date of 15 July 2014. Median follow up is 14.2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 24
months | 17.71 [17.710 to NA] — OS data are interim at data cutoff, with only 3 events in the study treatment phase (median follow-up 14.2 mos)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A serious AE is any AE occurring at any dose that: • Results in death; • Is life-threatening; • Requires or prolongs existing inpatient hospitalization; • Results in persistent or significant disability/incapacity; • Is a congenital anomaly/birth defect; • Constitutes an important medical event. The Investigator assessed the relationship of each AE to study drug and graded the severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0): Grade 1 = Mild (no limitation in activity or intervention required); Grade 2 = Moderate (some limitation in activity; no/minimal medical intervention required);-Grade 3 = Severe (marked limitation in activity; medical intervention required, hospitalization possible); Grade 4 = Life-threatening; Grade 5 = Death.
Time Frame: From first dose of study drug treatment through to 28 days after the last dose, until the data cut-off date of 15 July 2014; median treatment duration was 60 weeks
Population: Safety population includes all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lenalidomide Plus Dexamethasone
Number analyzed (Participants) | 26
participants
  Any adverse event | 26
  TEAE related to study drug | 25
  TEAE related to Lenalidomide | 25
  TEAE related to Dexamethasone | 20
  Grade 3-4 adverse event | 18
  Grade 3-4 adverse event related to any study drug | 15
  Grade 3-4 adverse event related to Lenalidomide | 15
  Grade 3-4 adverse event related to Dexamethasone | 4
  Serious TEAE | 11
  Serious TEAE related to any study drug | 8
  Serious TEAE related to Lenalidomide | 8
  Serious TEAE related to Dexamethasone | 3
  TEAE leading to discontinuation of either drug | 4
  TEAE leading to discontinuation of lenalidomide | 4
  TEAE leading to discontinuation of dexamethasone | 2
  Related TEAE discontinuation of either drug | 4
  Related TEAE discontinuation of lenalidomide | 4
  Related TEAE discontinuation of dexamethasone | 0

ADVERSE EVENTS:
Time Frame: From first dose of any study drug, through to 28 days after the last dose of the last study drugs received; until the data cut-off date of 14 July 2014. Maximum time on treatment was 89 weeks.
Groups:
- Lenalidomide Plus Dexamethasone: Lenalidomide: 25 mg oral lenalidomide once daily on Days 1 through 21 of each 28-day cycle
  Dexamethasone: 40 mg oral dexamethasone once daily on Days 1, 8, 15 and 22 of each 28-day cycle
Arm/Group | Lenalidomide Plus Dexamethasone
Serious Adverse Events (participants affected / at risk) | 11/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=26)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1
PNEUMONIA (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1
PRESYNCOPE (Nervous system disorders) | 1
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide Plus Dexamethasone (N=26)
RASH (Skin and subcutaneous tissue disorders) | 13
DRY SKIN (Skin and subcutaneous tissue disorders) | 5
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3
URTICARIA (Skin and subcutaneous tissue disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 8
STOMATITIS (Gastrointestinal disorders) | 3
DENTAL CARIES (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 2
VOMITING (Gastrointestinal disorders) | 2
OEDEMA PERIPHERAL (General disorders) | 6
MALAISE (General disorders) | 4
FACE OEDEMA (General disorders) | 2
NASOPHARYNGITIS (Infections and infestations) | 11
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
DYSGEUSIA (Nervous system disorders) | 4
ANAEMIA (Blood and lymphatic system disorders) | 8
NEUTROPENIA (Blood and lymphatic system disorders) | 7
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6
LEUKOPENIA (Blood and lymphatic system disorders) | 6
LYMPHOPENIA (Blood and lymphatic system disorders) | 4
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 3
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2
WEIGHT DECREASED (Investigations) | 2
INSOMNIA (Psychiatric disorders) | 6
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 4
HYPERTENSION (Vascular disorders) | 3
HYPOTENSION (Vascular disorders) | 2
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 3
HEAD INJURY (Injury, poisoning and procedural complications) | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 3
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
DIARRHOEA (Gastrointestinal disorders) | 2
GASTROENTERITIS (Infections and infestations) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
HYPOAESTHESIA (Nervous system disorders) | 2
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2
BLOOD CREATININE INCREASED (Investigations) | 2
BLOOD UREA INCREASED (Investigations) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
CONTUSION (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
CATARACT (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements varied; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.